CLINICAL TRIAL: NCT01343316
Title: Benefits of Post-Pyloric Feeding Tubes in Critically Ill Patients
Status: Terminated | Type: Observational
Why Stopped: lack of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Glenn Whitman, Associate Professor, Director of CVSICU and Adult Heart Transplant, Johns Hopkins University
Other Study IDs: NA_00041559
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Critical Illness
Keywords: Enteral Feeds; Supplemental Feeds; Transpyloric Tube; Nasogastric Tube
MeSH Terms: conditions — Critical Illness | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Transgastric tube: Nasogastric (NG tube)
  Interventions: Device: Transpyloric feeding tubes (Nasogastric Tube (NG tube), Tiger2, Syncro BlueTube)
- Transpyloric tube - Tiger2: Self-propelled by paristaltic waves of the stomach
  Interventions: Device: Transpyloric feeding tubes (Nasogastric Tube (NG tube), Tiger2, Syncro BlueTube)
- Transpyloric tube - Syncro BlueTube: Magnetically placed
  Interventions: Device: Transpyloric feeding tubes (Nasogastric Tube (NG tube), Tiger2, Syncro BlueTube)

INTERVENTIONS:
Device: Transpyloric feeding tubes (Nasogastric Tube (NG tube), Tiger2, Syncro BlueTube) — To determine the benefits of utilizing one type of transpyloric tube over another.
  Other Names: Nasogastric Tube (NG tube); Tiger2; Syncro BlueTube

SUMMARY:
The purpose of this study is to determine the benefit of feeding critically-ill patients beyond the stomach (post-pyloric). Furthermore, because of the advent of two new post-pyloric feeding tubes (Tiger 2 and Syncro BlueTube) designed to improve post-pyloric placement, the investigators will be evaluating the benefits of those two tubes as well.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the ICU who are deemed by the attending critical care physician to warrant tube feeds and expected to receive tube feeds for more than three days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients in the ICU setting
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine whether transpyloric feeds are superior to transgastric feeds with regard to ability to give calories and meet nutritional goals. | one year
  To determine the time to goal calories. To determine the number and qualitative aspect of tracheal aspirations. To determine the time to initiate tube feeds once the decision has been made to place a tube, the number of x-rays required for placement, the time required for placement, the number of times tube needs to be replaced.

SECONDARY OUTCOMES:
To determine the benefits of utilizing one type of transpyloric tube over another. One placed in the transpyloric position magnetically; the other propelled by peristalsis itself. | one year
  Benefits include shorter time to appropriate placement and quicker time to goal tube feed rate.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Whitman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Montejo JC, Minambres E, Bordeje L, Mesejo A, Acosta J, Heras A, Ferre M, Fernandez-Ortega F, Vaquerizo CI, Manzanedo R. Gastric residual volume during enteral nutrition in ICU patients: the REGANE study. Intensive Care Med. 2010 Aug;36(8):1386-93. doi: 10.1007/s00134-010-1856-y. Epub 2010 Mar 16. PMID 20232036
- [Background] Hsu CW, Sun SF, Lin SL, Kang SP, Chu KA, Lin CH, Huang HH. Duodenal versus gastric feeding in medical intensive care unit patients: a prospective, randomized, clinical study. Crit Care Med. 2009 Jun;37(6):1866-72. doi: 10.1097/CCM.0b013e31819ffcda. PMID 19384225
- [Background] Acosta-Escribano J, Fernandez-Vivas M, Grau Carmona T, Caturla-Such J, Garcia-Martinez M, Menendez-Mainer A, Solera-Suarez M, Sanchez-Paya J. Gastric versus transpyloric feeding in severe traumatic brain injury: a prospective, randomized trial. Intensive Care Med. 2010 Sep;36(9):1532-9. doi: 10.1007/s00134-010-1908-3. Epub 2010 May 22. PMID 20495781
- [Background] Heyland DK, Drover JW, MacDonald S, Novak F, Lam M. Effect of postpyloric feeding on gastroesophageal regurgitation and pulmonary microaspiration: results of a randomized controlled trial. Crit Care Med. 2001 Aug;29(8):1495-501. doi: 10.1097/00003246-200108000-00001. PMID 11505114
- [Background] Davies AR, Froomes PR, French CJ, Bellomo R, Gutteridge GA, Nyulasi I, Walker R, Sewell RB. Randomized comparison of nasojejunal and nasogastric feeding in critically ill patients. Crit Care Med. 2002 Mar;30(3):586-90. doi: 10.1097/00003246-200203000-00016. PMID 11990920